CLINICAL TRIAL: NCT03420976
Title: Pilot Study: Investigating a Novel Supplement-based Therapy for the Treatment of Small Intestinal Bacterial Overgrowth
Brief Title: Novel Supplement-based Therapy for the Treatment of Small Intestinal Bacterial Overgrowth
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PI no longer in practice.
Sponsor: Atrium Innovations (Industry)
Collaborators: Dr. Nathan Morris, MD (Unknown); Genova Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIBO-ATRGM2017
Record Dates: First submitted 2018-01-11; First posted 2018-02-05 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Small Intestinal Bacterial Overgrowth
Keywords: Small Intestinal Bacterial Overgrowth; SIBO

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Novel Supplement-based Therapy (Experimental): Low FODMAP diet + supplements outlined below:
  Product Name: Liver-G.I. Detox Active Ingredients: Alpha lipoic acid, n-acetyl-l-cystine, turmeric root extract, milk thistle seed extract, broccoli sprout concentrate, artichoke leaf extract, taurine, glycine, l-glutamine, l-methionine, and chlorella.
  Product Name: l-Glutamine Active Ingredients: l-glutamine
  Product Name: MicroDefense Active Ingredients: berberine sulfate, olive leaf extract, sweet wormwood, clove bud powder, and grapefruit seed and fruit extract.
  Product Name: A.C. Formulla II Active Ingredients: calcium and magnesium undecylenate, calcium and magnesium caprylate, bromelain, grapefruit seed and fruit extract, and berberine sulfate
  Product Name: Probiotic-5 (Pure Encapsulations) Active Ingredients: Probiotic blend
  Product Name: Digestive Enzymes Ultra with Betaine HCl Active Ingredients: Digestive enzyme blend and betaine HCl
  Interventions: Dietary Supplement: Novel Supplement Based Therapy

INTERVENTIONS:
Dietary Supplement: Novel Supplement Based Therapy — Supplements and Dosage:
  Detox Support: Liver-G.I. Detox BID for 30 days GI Support: L-Glutamine Powder 2 scoops QD for 35 days Microbial Balance: MicroDefense 1 capsule QD for 49 days Microbial Balance: A.C. Formula II 2 capsules BID for 49 days Probiotic: Probiotic-5 1 capsule QD for 49 days Digestive Enzymes: Digestive Enzymes Ultra with Betaine HCl As needed up to 6 longer term

SUMMARY:
Study Synopsis

This pilot study will determine the efficacy of a novel supplement protocol and low FODMAP diet for the treatment of small intestinal bacterial overgrowth (SIBO). The study will operate as a prospective, open label investigation, with an estimated sample size of 10 patients.

Patients diagnosed with SIBO by Dr. Nathan Morris, MD at Good Medicine Clinic (Oxford, Ohio) will be offered the opportunity to enroll in this study, if inclusion and exclusion criteria are met upon initial diagnosis. No control group will be assigned.

The diagnosis of SIBO will be determined via assessment of clinical symptoms and the results of a lactulose breath test. After administration of the supplement therapy and adherence to a low FODMAP diet (8 weeks), the lactulose breath test will be repeated and symptoms re-assessed by Dr. Morris. The post-treatment lactulose breath test and all supplements in the protocol will be provided free-of-charge to enrolled patients. In addition, enrolled patients will not be billed for the mid-treatment office visit. Patient and/or patient insurance will be responsible for all other expenses, including but not limited to the initial breath test, all other office visits and travel.

DETAILED DESCRIPTION:
Background

Small intestinal bacterial overgrowth (SIBO) is a category of gastrointestinal infection, characterized by an increased concentration (>100,000 CFU/mL proximal jejunal fluid) of bacteria in the small intestine. Symptoms of SIBO commonly afflict the gastrointestinal tract and include but are not limited to: abdominal pain, discomfort, bloating, cramping, flatulence, diarrhea, constipation, eructation, and low serum B12.

SIBO is believed to be severely under diagnosed and is associated with numerous comorbid conditions including irritable bowel syndrome, diabetes mellitus and hypothyroidism. Small-bowel aspiration (SBA) or breath tests are used to aid in the diagnosis of SIBO. Glucose or lactulose breath tests are more commonly performed, due to the cost and invasive nature of SBA.

Treatment of SIBO frequently consists of antibiotic therapy. Rifaxamin is a poorly absorbed antibiotic with bacteriocidal activity against enteropathogens that is widely prescribed for the treatment of SIBO. However, both patients and practitioners frequently turn to complementary and alternative treatment options, due to the adverse effects associated with antibiotic use and the recurrent nature of SIBO. In 2014, a retrospective study (Chedid et al.) found that the efficacy of a particular herbal therapy was comparable to Rifaxamin. However, both treatment options demonstrated a response rate of less than 50%. This investigation will test a more comprehensive, supplement-based therapy in hopes of achieving a greater response rate in patients diagnosed with SIBO.

Objectives

This investigation aims to determine the efficacy of a supplement protocol in combination with a low FODMAP diet for the treatment of SIBO.

Patient Selection

Patients diagnosed with SIBO at Dr. Morris' clinic will be offered the opportunity to enroll in this study as a theoretical treatment option for SIBO. Other treatment options will be discussed with the patient. Enrolled patients must satisfy the following inclusion and exclusion criteria:

Study Procedures

The supplement protocol is designed to take 8 weeks. Due to the delay in receiving and interpreting test results, the investigation, in its entirety, is estimated to take 12 weeks.

Visit -1 Dr. Morris will assess patient history and symptoms, at his facility in Oxford, Ohio. If suggestive of SIBO, a lactulose breath test will be prescribed. Additional testing may be performed, at the discretion of Dr. Morris, to aid in the initial diagnosis of the patient.

Visit 0 Dr. Morris will assess the results of the breath test and confirm or deny the diagnosis of SIBO. Treatment options for SIBO will be discussed, and the patient will be made aware of this investigation as a theoretical treatment option. Patient eligibility will be determined by completion of the the Patient Eligibility Checklist for each patient. All female patients will be asked to complete a urine pregnancy test to confirm pregnancy status. Eligible patients will be asked to review and sign the Informed Consent document. Carman Clark (Medical Assistant at Good Medicine) will be available to discuss patient consent and confidentiality. Enrolled patients will be asked to complete a baseline Medical Symptom Questionnaire. Afterwards, Ms. Clark will review the supplement therapy and low FODMAP diet. Patients will then be provided with all supplements necessary to complete the investigation. Patients will be asked to discontinue all other supplements during the study. No wash out period is required. Prescription medications, over-the-counter medications and/or supplements deemed medically necessary by the patient's primary care physician and/or Dr. Morris may be continued.

Visit 1 will occur approximately 4 weeks after the patient begins the supplement protocol. Patients will be asked to report their compliancy with the supplement protocol and low FODMAP diet and describe adverse effects. Patients will complete the Medical Symptom Questionnaire, be provided with the post-treatment lactulose breath test kit and instructed to perform the test within 2 weeks of completing the supplement therapy.

Visit 2 will occur after the results of the post-treatment breath test are available. Dr. Morris will interpret the results of the second breath test. Patients will again be asked to complete the Medical Symptom Questionnaire, report compliance with the supplement protocol and low FODMAP diet, and describe any adverse effects. Further treatment options will be discussed if necessary; follow-up treatment will be outside the scope of this investigation.

Risk/Safety Information

This study presents a risk in the form of adverse reactions to ingredients in the supplement therapy. Patient risk will be minimized by excluding patients who may respond poorly to the supplement therapy or testing procedures from the study, i.e., by abiding by the aforementioned patient enrollment exclusion criteria.

Monitoring/Reporting

Patients may report adverse events to Good Medicine during scheduled office visits or by phone during office hours. If serious or life-threatening side effects arise, patients are instructed to call 911. Possible side effects include but are not limited to: diarrhea, constipation, nausea, vomiting, bloating or headache. When necessary, Dr. Morris or Ms. Clark will communicate with patients outside the office by phone. Medical guidance will be provided as necessary. Adverse events will be recorded in confidential patient files.

Study Oversight

This study will be terminated if one-half or more of enrolled patients withdraw due to adverse events. Dr. Morris and Dr. Kelly Heim (Senior Director, Scientific Affairs at Atrium Innovations) will monitor, determine the need for and facilitate the termination of the study. Direct access to study related data will be made available for monitoring, auditing, IRB review and regulatory inspection.

ELIGIBILITY:
Inclusion Criteria:

A positive diagnosis of SIBO, which will be defined by:

1. presentation of the aforementioned symptoms and
2. positive results of a lactulose breast test. Positive breath test results will be defined as an increase in hydrogen of 20 ppm or more and/or an increase in methane of 12 ppm or more compared to baseline by 90 minutes.

Exclusion Criteria:

1. Use of prescription antibiotics or antifungals within the past 4 weeks.
2. Younger than 18 or older than 85 years of age.
3. Pregnant or breastfeeding.
4. Major drug-supplement interactions between essential medication and the proposed supplement therapy.
5. A known allergy to one or more of the ingredients in the supplement therapy.
6. Has been diagnosed and treated for SIBO within the past 6 months.
7. Has undergone a colonoscopy or barium enema within the past 4 weeks.
8. Has an allergy to lactulose. 9) Has diabetes mellitus.

Ages: 19 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2019-01-30 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
Lactulose Breath Test | 8 weeks
  Clinically and/or statistically significant reduction in hydrogen and methane levels following lactulose ingestion

SECONDARY OUTCOMES:
Symptom Survey | 8 weeks
  Patient reported remission or improvement of SIBO-related symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Morris, MD, Principal Investigator — Good Medicine
Locations (1):
- Good Medicine, Oxford, Ohio, United States

DOCUMENTS (1):
  • Study Protocol (2017-05-03): https://cdn.clinicaltrials.gov/large-docs/76/NCT03420976/Prot_000.pdf